CLINICAL TRIAL: NCT00915889
Title: Cervical Cancer Survivorship Among African-, European-, and Latina-American Survivors
Brief Title: Psychosocial Support for African-American, Latina-American, or European-American Cervical Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06081; P30CA033572 (NIH); CHNMC-06081; CDR0000642406 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Cancer Survivor; Cervical Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; stage IA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; cancer survivor
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Counseling; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Active Comparator): Patients receive a survivorship booklet in the mail that contains information about cervical cancer. Patients then receive a follow-up telephone call at 3 months to clarify any issues relevant to the survivorship booklet.
  Interventions: Other: questionnaire administration
- Group II (Experimental): Patients are randomly assigned to receive either 6 or 8 weekly telephone sessions that address managing medical issues, health education, and cancer resources; balancing emotions and managing stress; coping skills and problem solving; family and social concerns; relational, intimacy, and sexual concerns; and financial and employment concerns. Patients also receive a survivorship booklet as in group I.
  Interventions: Behavioral: telephone-based intervention; Other: counseling intervention; Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Procedure: psychosocial assessment and care

INTERVENTIONS:
Behavioral: telephone-based intervention — Either 6 or 8 telephone educational sessions
  Arms: Group II
Other: counseling intervention — counseling and communications studies
  Arms: Group II
Other: questionnaire administration — Ancillary studies
Other: study of socioeconomic and demographic variables — Ancillary Studies
  Arms: Group II
Procedure: psychosocial assessment and care — 6 weeks or 8 weeks of psychoeducational telephone sessions
  Arms: Group II

SUMMARY:
RATIONALE: Telephone counseling may help reduce depression and anxiety and improve the well-being and quality of life of cervical cancer survivors.

PURPOSE: This randomized clinical trial is studying how well psychosocial support works in African-American, Latina-American, or European-American cervical cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES: I. To evaluate the utility of the 6 telephone sessions (low intensity: LiTx) and 8 telephone sessions (high intensity: HiTx) plus Survivorship Booklet designed to educate and improve awareness of the physical and psychological impact of cancer and increase knowledge of appropriate medical and psychosocial resources for women with cervical cancer. II. To evaluate the utility of the telephone sessions (LiTx and HiTx) designed to improve psychological functioning (decrease depression and anxiety) of women with cervical cancer. III. To evaluate the utility of the telephone sessions (LiTx and HiTx) designed to improve social functioning (family support and communication).

OUTLINE: Patients are clinically assigned to 1 of 2 groups. GROUP I: Patients receive a survivorship booklet in the mail that contains information about cervical cancer. Patients then receive a follow-up telephone call at 3 months to clarify any issues relevant to the survivorship booklet. GROUP II: Patients are randomly assigned to receive either 6 or 8 weekly telephone sessions that address managing medical issues, health education, and cancer resources; balancing emotions and managing stress; coping skills and problem solving; family and social concerns; relational, intimacy, and sexual concerns; and financial and employment concerns. Patients also receive a survivorship booklet as in group I.

ELIGIBILITY:
Inclusion Criteria: Within 6 months to 3 years of a cervical cancer diagnosis Diagnosed with stages 1-3 invasive cervical cancer Not diagnosed with another type of cancer No other major disabling medical or psychiatric condition Survivors within 6 months to 3 years post diagnosis are included Participants must be able to read and/or speak either English or Spanish Women will not be excluded based on the type of treatment received for their cervical cancer or a history of diagnosis of mild depression or anxiety Exclusion Criteria: Women with metastatic disease Women with major medical conditions (e.g., stroke and degenerative illness) Survivors with moderate to severe depression or anxiety Asian participants Stage 0 disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2006-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Utility of a psychosocial intervention in educating and improving awareness of the physical and psychological impact of cancer and in increasing knowledge about appropriate medical and psychosocial resources for cervical cancer survivors | 12 months after study initiation
Utility of a psychosocial intervention in improving psychological functioning (i.e., decreasing depression and anxiety) among cervical cancer survivors | 12 months after study initiation
Utility of a psychosocial intervention in improving social functioning (i.e., family support and communication) among cervical cancer survivors | 12 months after study initiation

CONTACTS AND LOCATIONS:
Overall Officials: Kimlin Ashing-Giwa, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States